CLINICAL TRIAL: NCT03567187
Title: Cryoneurolysis for Improvements in Pain, Activities of Daily Living and Quality of Life in Patients With Ankle Osteoarthritis
Brief Title: Cryoneurolysis for Improvements in Pain, ADL and QOL in Patients With Ankle Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Neil Segal, MD, MS, Professor, University of Kansas Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142298
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Ankle Osteoarthritis
Keywords: Cryoneurolysis; iovera; Superficial nerves treatment; Deep Fibular Nerve

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Iovera (Experimental): The iovera° device consists of a reusable, portable hand-piece, along with a single-patient use sterile smart Tip (cryoprobe) and disposable nitrous oxide (N2O) cartridges (cryogen). The smart tip is composed of closed-tip stainless steel needles, thereby fully enclosing the cryogen. There are 2 types of smart tips that will be utilized during this study, depending on the depth of the nerves being treated. The shorter smart tip comes in 2 variants - three X 6.9 mm or 8.9 mm, 27-gauge needles, with an attached skin warmer to prevent damage to the underlying skin. The longer smart tip also comes in 2 variants - 55 mm 22-gauge needle or a 90 mm 20G needle.
  The effect is by initiation of a cooling cycle, by fully inserting the smart tip into the procedure site and activating the cryogen flow. As the gas travels through the length of the needle, an ice ball develops around the needle freezing the surrounding tissue.
  Interventions: Device: iovera

INTERVENTIONS:
Device: iovera — The iovera° device is 510(k)-cleared (K133453 and K161835) and is used to form a precisely controlled, sub-dermal cold zone of -20 to -88.5 degrees Celsius to temporarily disrupt peripheral nerve function, ultimately blocking pain. It is not indicated for the treatment of central nervous system tissue.

SUMMARY:
This will be an open-label trial to describe the effects of cryoneurolysis with iovera° on symptom relief in patients with painful Kellgren-Lawrence (KL) grade 2-4 ankle osteoarthritis (OA). The Foot and Ankle Outcome Score (FAOS) subscales will be used to assess outcomes at 6, 12 and 24 weeks after treatment.

DETAILED DESCRIPTION:
The aim of this study is to assess clinically significant long-term symptomatic relief with cryoneurolysis in people with unilateral ankle osteoarthritis (OA). The investigators will treat 1) the Superficial Fibular Nerve (SFN), Sural Nerve (SN) and Saphenous Nerve and/or 2) the Deep Fibular Nerve (DFN) with cryoneurolysis using the iovera° device. The primary study endpoint, clinically significant improvement in pain 12 weeks after each treatment, will be assessed using the FAOS pain subscale. If a participant is a non-responder (<20% improvement in pain within the 12 weeks following baseline), then the other treatment will be offered (e.g. if start with superficial group, then offer the DFN).

The secondary outcomes will be improvement in quality of life (FAOS-QoL), activities of daily living (FAOS-ADL) and Numerical Rating Scale (NRS) for pain.

The tertiary outcome will be improvement in physical performance measures (40m fast-paced walking test, standing balance test).

ELIGIBILITY:
Inclusion Criteria:

* Participation in an institutional review board-approved informed consent process, culminating in providing written consent.
* Willingness and ability to comply with the study procedures, visit schedules and ability to follow verbal and written instructions.
* Male or female over 18 years of age.
* Currently Kellgren-Lawrence (KL) Grade 2, 3 or 4 in the ankle based on X-ray (weight-bearing mortise views with 20° internal rotation) or weight-bearing CT scan of the ankles.
* Limited by unilateral ankle pain, rated on a Numerical Rating Scale for pain severity as ≥5 on most days over the last month.
* Foot and ankle outcome score (FAOS) of < 75 in at least 1 category.
* Body mass index (BMI) ≤ 50 kg/m2
* Ambulatory
* Willingness to abstain from the use of protocol-restricted medications during the study and also willing to abstain from use of analgesics other than acetaminophen 1 week prior to beginning of the study.
* Has undergone at least one prior conservative osteoarthritis treatment (e.g. physical therapy, analgesics).

Exclusion Criteria:

* Baseline knee, hip, spine or other limitations that affect walking ability to a greater extent than the ankle.
* Cryoglobulinemia, paroxysmal cold hemoglobinuria, Raynaud's disease, cold urticaria.
* Clinical signs or symptoms of active or recurrent infection in the index ankle joint or overlying skin.
* Intra-articular, intravenous or intramuscular corticosteroid (investigational or marketed) within 3 months of screening
* Oral corticosteroids (investigational or marketed) within 2 weeks of screening (unless on a chronic stable dose for ≥3 months prior to enrollment).
* Women who are pregnant (due to potential for the change in body mass and distribution to alter ankle symptoms over the period of follow-up).
* Any condition other than OA of the ankle joint which, in the opinion of the investigators, affects their ability to ambulate to a sufficient degree to interfere with the assessment of the safety and treatment effects of the study injection.
* Arthroscopy or open surgery of the ankle joint within 6 months of screening.
* Planned/anticipated surgery of the index ankle joint during the 6-month study period.
* Any clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the investigator, could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study injection.
* Skin breakdown at the ankle joint where the injection is planned to take place.
* Participated in any investigational drug or device trial within 30 days prior to screening or concurrent participation in another research study that could complicate interpretation of the findings of either study.
* Current consumption of more than 14 alcoholic drinks per week.
* Patients with diffuse pain conditions (Complex pain - diffuse or confounding pain, fibromyalgia, etc.).
* Known altered nerve anatomy or physiology (e.g. neuropathy) at the target, such as due to a congenital, traumatic or surgical cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward ST, Williams PL, Purkayastha S. Intra-articular corticosteroid injections in the foot and ankle: a prospective 1-year follow-up investigation. J Foot Ankle Surg. 2008 Mar-Apr;47(2):138-44. doi: 10.1053/j.jfas.2007.12.007. PMID 18312921
- [Background] Valderrabano V, Horisberger M, Russell I, Dougall H, Hintermann B. Etiology of ankle osteoarthritis. Clin Orthop Relat Res. 2009 Jul;467(7):1800-6. doi: 10.1007/s11999-008-0543-6. Epub 2008 Oct 2. PMID 18830791
- [Background] Repetto I, Biti B, Cerruti P, Trentini R, Felli L. Conservative Treatment of Ankle Osteoarthritis: Can Platelet-Rich Plasma Effectively Postpone Surgery? J Foot Ankle Surg. 2017 Mar-Apr;56(2):362-365. doi: 10.1053/j.jfas.2016.11.015. PMID 28231968
- [Background] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882
- [Background] Evans PJ, Lloyd JW, Green CJ. Cryoanalgesia: the response to alterations in freeze cycle and temperature. Br J Anaesth. 1981 Nov;53(11):1121-7. doi: 10.1093/bja/53.11.1121. PMID 7326160
- [Background] Golightly YM, Devellis RF, Nelson AE, Hannan MT, Lohmander LS, Renner JB, Jordan JM. Psychometric properties of the foot and ankle outcome score in a community-based study of adults with and without osteoarthritis. Arthritis Care Res (Hoboken). 2014 Mar;66(3):395-403. doi: 10.1002/acr.22162. PMID 24023029
- [Background] Mani SB, Do H, Vulcano E, Hogan MV, Lyman S, Deland JT, Ellis SJ. Evaluation of the foot and ankle outcome score in patients with osteoarthritis of the ankle. Bone Joint J. 2015 May;97-B(5):662-7. doi: 10.1302/0301-620X.97B5.33940. PMID 25922461
- [Background] Holzer N, Salvo D, Marijnissen AC, Vincken KL, Ahmad AC, Serra E, Hoffmeyer P, Stern R, Lubbeke A, Assal M. Radiographic evaluation of posttraumatic osteoarthritis of the ankle: the Kellgren-Lawrence scale is reliable and correlates with clinical symptoms. Osteoarthritis Cartilage. 2015 Mar;23(3):363-9. doi: 10.1016/j.joca.2014.11.010. Epub 2014 Nov 15. PMID 25463444
- [Background] Roos EM, Brandsson S, Karlsson J. Validation of the foot and ankle outcome score for ankle ligament reconstruction. Foot Ankle Int. 2001 Oct;22(10):788-94. doi: 10.1177/107110070102201004. PMID 11642530
- [Background] Hunt KJ, Hurwit D. Use of patient-reported outcome measures in foot and ankle research. J Bone Joint Surg Am. 2013 Aug 21;95(16):e118(1-9). doi: 10.2106/JBJS.L.01476. PMID 23965711
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] McDaniel G, Renner JB, Sloane R, Kraus VB. Association of knee and ankle osteoarthritis with physical performance. Osteoarthritis Cartilage. 2011 Jun;19(6):634-8. doi: 10.1016/j.joca.2011.01.016. Epub 2011 Feb 19. PMID 21310252
- [Result] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-three potentially eligible participants were screened. Of these two were found by radiographs or weight-bearing CT (WBCT) scan to not have tibiotalar osteoarthritis (KL=0) and were excluded. In addition, one participant was excluded due to an unstable ankle that resulted in bracing and opioid therapy. Subsequently, 40 participants with unilateral painful ankle OA were recruited.
Groups:
- Iovera: The iovera° device consists of a reusable, portable hand-piece, along with a single-patient use sterile smart Tip (cryoprobe) and disposable nitrous oxide (N2O) cartridges (cryogen). The smart tip is composed of closed-tip stainless steel needles, thereby fully enclosing the cryogen. There are 2 types of smart tips that will be utilized during this study, depending on the depth of the nerves being treated. The shorter smart tip comes in 2 variants - three X 6.9 mm or 8.9 mm, 27-gauge needles, with an attached skin warmer to prevent damage to the underlying skin. The longer smart tip also comes in 2 variants - 55 mm 22-gauge needle or a 90 mm 20G needle.
  The effect is by initiation of a cooling cycle, by fully inserting the smart tip into the procedure site and activating the cryogen flow. As the gas travels through the length of the needle, an ice ball develops around the needle freezing the surrounding tissue.
  iovera: The iovera° device is 510(k)-cleared (K133453 and K161835) and is used to form a precisely controlled, sub-dermal cold zone of -20 to -88.5 degrees Celsius to temporarily disrupt peripheral nerve function, ultimately blocking pain. It is not indicated for the treatment of central nervous system tissue.
Period: Overall Study
Arm/Group | Iovera
Started | 40
Completed | 22
Not Completed | 18
Not completed — Lost to Follow-up | 18

BASELINE CHARACTERISTICS:
Population: Forty-three potentially eligible participants were screened. Of these, two were found by radiographs or weight-bearing CT (WBCT) scan to not have tibiotalar osteoarthritis (KL = 0) and were excluded. In addition, one participant was excluded due to an unstable ankle that resulted in bracing and opioid. Subsequently, 40 participants with unilateral painful ankle OA were recruited.
  therapy. Subsequently, 40 participants with unilateral painful ankle OA were recruited.
Arm/Group | Iovera
Number analyzed (Participants) | 40
Age, Continuous [Least Squares Mean (Standard Deviation); unit: years] | 63.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 40
NRS Pain Score [Mean (Standard Deviation); unit: units on a scale] — Pain in past 7 days
  units on a scale | 6.3 (1.6)
FAOS-Pain [Mean (Standard Deviation); unit: units on a scale] | 43.1 (14.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.7 (6.8)
Index ankle joint, n (% right ) [Count of Participants; unit: Participants] | 27
FAOS-ADL [Mean (Standard Deviation); unit: units on a scale] | 53.3 (16.4)
FAOS-QOL [Mean (Standard Deviation); unit: units on a scale] | 22.0 (16.9)
40-meter fast-paced walking test [Mean (Standard Deviation); unit: sec] | 32.8 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: FAOS - PAIN
Description: FAOS-Pain is a subscale of the Foot and ankle outcome score (FAOS) which is a self-reported outcome score.The sub scale ranges from 0 to 100 where higher values represents a better outcome.
Time Frame: Change between baseline/screening and 12-weeks following treatment
Population: Twenty seven eligible participants completed 12-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 27
score on a scale | 20.8 (4.5)

2. Secondary Outcome: NRS Pain Over Prior 7 Days
Description: The Numeric Rating Scale (NRS) is a numeric scale to rates the pain from 0 (no pain) to 10 (worst pain).
Time Frame: change between baseline/screening and 6-weeks following treatment
Population: Thirty five eligible participants completed 6-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 35
score on a scale | -2.7 (0.5)

3. Secondary Outcome: FAOS - ADL(Activity of Daily Living)
Description: FAOS - ADL(Activity of daily living) is a subscale of the Foot and ankle outcome score (FAOS) which is a self-reported outcome score. It is similar to the KOOS - ADL components.The sub scale ranges from 0 to 100 where higher values represents a better outcome.
Time Frame: change between baseline/screening and 12-weeks following treatment
Population: Twenty seven eligible participants completed 12-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 27
score on a scale | 18.1 (4.9)

4. Secondary Outcome: FAOS - ADL(Activity of Daily Living)
Description: as for outcome 3
Time Frame: change between baseline/screening and 6-weeks following treatment
Population: Thirty five eligible participants completed 6-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 35
score on a scale | 16.6 (4.3)

5. Secondary Outcome: FAOS - ADL(Activity of Daily Living)
Description: as for outcome 3
Time Frame: change between baseline/screening and 24-weeks following treatment
Population: Twenty two eligible participants completed 24-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 22
score on a scale | 20.1 (4.1)

6. Secondary Outcome: FAOS-QoL(Quality of Life)
Description: FAOS-QoL(Quality of life) is a subscale of the Foot and ankle outcome score (FAOS) which is a self-reported outcome score. It is similar to the KOOS - QoL components.The sub scale ranges from 0 to 100 where higher values represents a better outcome.
Time Frame: change between baseline/screening and 12-weeks following treatment
Population: Twenty seven eligible participants completed 12-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 27
score on a scale | 19.9 (5.3)

7. Secondary Outcome: FAOS-QoL(Quality of Life)
Description: as for outcome 6
Time Frame: change between baseline/screening and 6-weeks following treatment
Population: Thirty five eligible participants completed 6-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 35
score on a scale | 22.4 (4.4)

8. Secondary Outcome: FAOS-QoL(Quality of Life)
Description: as for outcome 6
Time Frame: change between baseline/screening and 24-weeks following treatment
Population: Twenty two eligible participants completed 24-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 22
score on a scale | 25.4 (4.8)

9. Secondary Outcome: FAOS - PAIN
Description: as for outcome 1
Time Frame: change between baseline/screening and 6-weeks following treatment
Population: Thirty five eligible participants completed 6-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 35
score on a scale | 17.4 (4.1)

10. Secondary Outcome: FAOS - PAIN
Description: as for outcome 1
Time Frame: change between baseline/screening and 24-weeks following treatment
Population: Twenty two eligible participants completed 24-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 22
score on a scale | 21.7 (4.3)

11. Secondary Outcome: NRS Pain Over Prior 7 Days
Description: The Numeric Rating Scale (NRS) is a numeric scale to rates the pain from 0 (no pain) to 10 (worst pain).
Time Frame: change between baseline/screening and 24-weeks following treatment
Population: Twenty two eligible participants completed 24-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 22
score on a scale | -2.8 (0.5)

12. Secondary Outcome: NRS Pain Over Prior 7 Days
Description: The Numeric Rating Scale (NRS) is a numeric scale to rates the pain from 0 (no pain) to 10 (worst pain).
Time Frame: change between baseline/screening and 12-weeks following treatment
Population: Twenty seven eligible participants completed 12-weeks follow-up treatment
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Iovera
Number analyzed (Participants) | 27
score on a scale | -2.6 (0.6)

13. Other Pre Specified Outcome: Change in 40m Fast Paced Walking Test (40m FPWT) Time Between Baseline/Screening and 6-weeks Following Treatment
Description: The 40-meter walk test is one of the three OARSI (Osteoarthritis Research Society International) recommended minimal core set of performance-based outcome measures in OA research and clinical practice.The 40m FPWT will take approximately 2 minutes for each subject to complete.
Time Frame: change between baseline/screening and 6-weeks following treatment
Population: Thirty five eligible participants completed 6-weeks follow-up treatment
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Iovera
Number analyzed (Participants) | 35
seconds | -0.1 (2.3)

14. Other Pre Specified Outcome: Change in 40m Fast Paced Walking Test (40m FPWT) Time Between Baseline/Screening and 12-weeks Following Treatment
Description: as for outcome 13
Time Frame: change between baseline/screening and 12-weeks following treatment
Population: Twenty seven eligible participants completed 12-weeks follow-up treatment
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Iovera
Number analyzed (Participants) | 27
seconds | -1.2 (2.2)

15. Other Pre Specified Outcome: Change in 40m Fast Paced Walking Test (40m FPWT) Time Between Baseline/Screening and 24-weeks Following Treatment
Description: as for outcome 13
Time Frame: change between baseline/screening and 24-weeks following treatment
Population: Twenty two eligible participants completed 24-weeks follow-up treatment
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Iovera
Number analyzed (Participants) | 22
seconds | -1.8 (2.6)

ADVERSE EVENTS:
Time Frame: All participants were followed for up to 24-weeks post cryoneurolysis treatment. Demographic and clinical characteristics for all participants were captured at baseline, 3, 6, 9, 12, 18 and 24-weeks follow-up.
Description: Over the 24-week follow-up period following cryoneurolysis treatment, 19 participants reported a total of 42 adverse events. Of these, 2 were deemed to be unrelated to the intervention, 4 unlikely related, 18 possibly related, 14 probably related and 5 definitely related. The most frequently reported adverse events were index ankle arthralgia and paraesthesia. There were no serious adverse events.
Arm/Group | Iovera
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 19/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iovera (N=40)
arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14)
Bruising (Vascular disorders) | 2 (2)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
fall (General disorders) | 2 (2)
localized edema (Blood and lymphatic system disorders) | 5 (5)
muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (3)
pain ( 1st web space) (Musculoskeletal and connective tissue disorders) | 1 (1)
paraesthesia (Nervous system disorders) | 11 (11)
pruritus (Immune system disorders) | 1 (1)
skin disorder - other (lump) (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/87/NCT03567187/Prot_SAP_000.pdf